CLINICAL TRIAL: NCT07183683
Title: Electrical Versus Manual Stimulation of Acupuncture Points in Female Patients With Multiple Sclerosis and Neurogenic Bladder Dysfunction - A Pragmatic, Exploratory, Three-Arm, Randomized Controlled Trial Using a Mixed Methods Approach
Brief Title: Stimulation of Acupuncture Points in Female Patients With Multiple Sclerosis and Neurogenic Bladder Dysfunction
Acronym: ACULUTS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Benno Brinkhaus, Professor Dr. Benno Brinkhaus, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACULUTS-MS KVC; KVC 01/143/2024 (Other Grant/Funding Number: Karl and Veronica Carstens foundation)
Record Dates: First submitted 2025-09-11; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Neurogenic Bladder Dysfunction
Keywords: multiple sclerosis; urinary bladder dysfunction; electrical stimulation; acupressure; acupuncture; posterior tibial nerve
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- group 1: electrical stimulation of acupuncture points plus routine care (Experimental): Intervention is electrical stimulation of two acupuncture points at the inner ankle of the foot over the posterior tibialis nerve, stimulation twice daily over 5 weeks
  Interventions: Device: group 1: electrical stimulation of acupuncture points plus routine care
- group 2: acupressure plus routine care (Experimental): manual stimulation of the same two acupressure points over the inner ankle, stimulation twice daily over 5 weeks
  Interventions: Other: group 2: acupressure plus routine care
- group 3: routine care alone (No Intervention): waiting list control

INTERVENTIONS:
Device: group 1: electrical stimulation of acupuncture points plus routine care — The acupuncture points Spleen 6 and Kidney 3 will be stimulated twice daily with a up to 30min electrical stimulation per foot with 10Hz and an intensity up to individual tolerance level.
  Other Names: posterior tibial nerve stimulation
  Arms: group 1: electrical stimulation of acupuncture points plus routine care
Other: group 2: acupressure plus routine care — The acupuncture points Spleen 6 and Kidney 3 will be stimulated twice daily with a up to 30min massage per foot
  Arms: group 2: acupressure plus routine care

SUMMARY:
Electrical vs. manual stimulation: The study compares two types of acupuncture - one using mild electrical currents and one using just manual no-needle techniques in the treatment of urinary bladder disfunction.

The study focuses on women diagnosed with multiple sclerosis (MS) who also have neurogenic bladder dysfunction - a condition where the bladder doesn't work properly due to nerve damage.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the feasibility, therapeutic effects, and safety of (A) electrical stimulation of acupuncture points (using a TENS device) in addition to routine care, and (B) manual stimulation of acupuncture points (using acupressure) in addition to routine care, compared to (C) routine care alone (control group), in female patients with multiple sclerosis (MS) and neurogenic bladder dysfunction.

Key outcome parameters include symptoms of neurogenic bladder dysfunction assessed using standardized patient-reported outcome measures.

Moreover, a qualitative substudy will be conducted to explore the subjectively perceived effects of the study interventions and the overall feasibility of the study. This will be carried out through semi-structured interviews and analyzed using qualitative research methodology.

ELIGIBILITY:
Inclusion Criteria:

* Female patients, aged 18-60 years, with relapsing-remitting multiple sclerosis (RRMS) and an Expanded Disability Status Scale (EDSS) score ≤ 6
* Stable immunomodulatory MS therapy for at least 3 months prior to enrollment
* Presence of at least 3 out of the following 6 criteria indicative of overactive bladder dysfunction: urgency, daytime urinary frequency >10 times, nocturia >1 time per night, post-void dribbling, incontinence, or delayed initiation of micturition
* Participants must be willing and cognitively and linguistically capable of adhering to the study protocol, performing the study interventions, and completing the required study documentation
* Capacity to provide informed consent, and provision of written consent for both written and electronic data collection and participation in the study

Exclusion Criteria:

* Acute MS relapse within the last 3 months prior to individual study entry
* Planned change in immunomodulatory therapy during the study period
* Current need for regular self-catheterization (more than twice per week)
* Clinically relevant post-void residual volume, confirmed by ultrasound (>100 mL or >40% of pre-void volume)
* Current or past history of bladder cancer
* Implanted defibrillator or other pacemaker
* Urogenital causes of bladder dysfunction, such as stress urinary incontinence or bladder prolapse
* Spinal trauma within 5 years prior to study entry or any other pre-existing central nervous system disorders (e.g., stroke, Parkinson's disease), or history of pelvic, spinal, or bladder surgery
* Acute urinary tract infection at the time of screening or within the previous 4 weeks
* Urolithiasis or urogenital tumors within the past 6 months
* Previous electrical posterior tibial nerve stimulation (TNS), acupuncture, or acupressure in the same anatomical region within 3 months prior to study entry
* Regular pelvic floor training (more than twice per week) in the past 6 weeks or planned during the study period
* Planned participation in another interventional clinical trial during the study period
* Open wounds, edema, or lymphedema in the lower leg that may interfere with local intervention
* Other serious pre-existing conditions (e.g., active cancer, heart failure, epilepsy, etc.) that contraindicate participation in the study
* Obesity, defined as BMI > 30
* Pregnancy or breastfeeding

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Incontinence Questionnaire Overactive Bladder (ICIQ-OAB) | weeks 5 and 10 after the start of the intervention
  Bladder function scoring 0-16, higher values mean worse outcome

SECONDARY OUTCOMES:
Incontinence Quality of Life Measure (I-QoL) | weeks 5 and 10 after the start of the intervention
  Disease-specific quality of life, scoring 1-110 , the higher the values the better
Patient's Global Impression of Change (PGIC) | weeks 5 and 10 after the start of the intervention
  Subjective improvement of bladder dysfunction since start of the study, onedimenional scale with seven grades ranging from 'very much worse' to 'very much improved'
3-day voiding diary | weeks 5 and 10 after the start of the intervention
  Objective voiding parameters, including mean voiding frequency and average fluid intake to urine output ratio, assessing daytime urination frequency
100mm Visual Analogue pain Scale (VAS) for last menstruation | at weeks 5 and 10
  Pain during the most recent menstruation ranging from 0: no pain to 100: maximum pain

OTHER OUTCOMES:
rate of rescue medication | between weeks 1 and 5 and at week 10
  rate of use of rescue medication (e.g., anticholinergics) and self-catheterization during trial participation
rate of adverse events | from week 1 to 10
  the Safety of intervention will be assessed by recording the rate of adverse events and identification of adverse reactions

CONTACTS AND LOCATIONS:
Locations (1):
- Department for integrative medicine and prevention, Institute for social medicine, epidemiology and health economics, Charité university medicine Berlin, Berlin, State of Berlin, Germany

IPD SHARING:
Plan to Share IPD: Yes
under reasonable request
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: from 31.12.2027- 31.12.2032

REFERENCES:
- [Background] Al Dandan HB, Coote S, McClurg D. Prevalence of Lower Urinary Tract Symptoms in People with Multiple Sclerosis: A Systematic Review and Meta-analysis. Int J MS Care. 2020 Mar-Apr;22(2):91-99. doi: 10.7224/1537-2073.2019-030. PMID 32410904
- [Background] Chang KK, Wong TK, Wong TH, Leung AW, Chung JW. Effect of acupressure in treating urodynamic stress incontinence: a randomized controlled trial. Am J Chin Med. 2011;39(6):1139-59. doi: 10.1142/S0192415X11009469. PMID 22083987
- [Background] Marzouk MH, Darwish MH, El-Tamawy MS, Morsy S, Abbas RL, Ali AS. Posterior tibial nerve stimulation as a neuromodulation therapy in treatment of neurogenic overactive bladder in multiple sclerosis: A prospective randomized controlled study. Mult Scler Relat Disord. 2022 Dec;68:104252. doi: 10.1016/j.msard.2022.104252. Epub 2022 Oct 17. PMID 36274285
- [Background] Guitynavard F, Mirmosayyeb O, Razavi ERV, Hosseini M, Hosseinabadi AM, Ghajarzadeh M, Azadvari M. Percutaneous posterior tibial nerve stimulation (PTNS) for lower urinary tract symptoms (LUTSs) treatment in patients with multiple sclerosis (MS): A systematic review and meta-analysis. Mult Scler Relat Disord. 2022 Feb;58:103392. doi: 10.1016/j.msard.2021.103392. Epub 2021 Nov 10. PMID 35216773